CLINICAL TRIAL: NCT00190372
Title: Contribution of a Psycho-Educational Program of Help to Help in the Pharmacological Assumption of Responsibility of the Disease of Alzheimer
Brief Title: AIDMA: A Psycho-educational Program Designed to Support and Train Carers of Alzheimer's Disease (AD) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Amel OUSLIMANI, Department of Clinical Research of developpement
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: P030437
Record Dates: First submitted 2005-09-14; First posted 2005-09-19 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2007-03

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease training programme; educational programme caregivers carers dementia treatment; Dementia Cognitive disorder
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Other)
  Interventions: Behavioral: Controlled diet; Behavioral: Self-hypnotic relaxation

INTERVENTIONS:
Behavioral: Controlled diet — Controlled diet
Behavioral: Self-hypnotic relaxation — Self-hypnotic relaxation

SUMMARY:
The aim of the project is to demonstrate that a psycho-educational programme designed to support and train carers of Alzheimer's disease (AD) patients induces a significantly higher benefit than anticholinesterase drug treatment alone or associated to memantine treatment. This training programme focuses on the explanation/description of behavioral, cognitive and functional disorders induced by the disease, as well as principles of cognitive and psycho-social stimulation of the patients in daily life.

DETAILED DESCRIPTION:
Context: Research showing the benefit of a combined approach including specific antidementia drugs and psycho-educational programmes for caregivers in the caring of Alzheimer's disease patients is still lacking. We venture the hypothesis that combined treatment including a specific antidementia drug for the AD patient and a psycho-educational programme for the caregivers has a larger benefit for both the patient and the caregiver on psychological, behavioural, and cognitive parameters.

Main objective: to demonstrate that a psycho-educational programme designed to support and train carers of Alzheimer's disease (AD) patients induces a significantly higher benefit than anticholinesterase drug treatment alone or associated to memantine treatment.

Secondary objective: identify patterns of responders and non-responders (taking into account cognitive, psychological parameters).

Methodology: national multicentric, randomized trial, single blinded, with 2 parallel groups of 120 patients and 120 caregivers trained for a 3 month period with 3 assessments: before, just after and 3 months after the training period. Patients and caregivers are recruited (according to exclusion and inclusion criteria) and followed up in memory centers participating in the trial.

Evaluation criteria:

Primary criteria for the patient: DAD scale (Disability Assessment for Dementia).

Secondary evaluation criteria - for the patient: NPI and ADAS-Cog; for the caregiver: ZARIT scale, Questionnaire of feeling of competency, Montgomery and Asberg Depression Rating Scale (MADRS), Geriatric Depression Scale (GDS).

Statistical analysis by the department of biostatistics and medical computing of the Hospital Cochin will be performed.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* AD outpatients
* Stable pharmacological treatment
* Mini-Mental State Examination (MMSE) [10 -28]
* Age [60-90]
* Informed consent

Caregivers:

* Reliability
* Motivation
* Psychological disorder related to patient's disease
* Need for information or help
* Informed consent

Exclusion Criteria:

Patients:

* Other dementia
* Severe general disease
* No reliable caregiver

Caregivers:

* Physical or mental disease incompatible with patient's management
* Impossibility to participate in the educational program
* Absence of anxiety-depression
* Psychotherapy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2004-10; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
DAD scale (Disability Assessment for Dementia) | at 6 months

SECONDARY OUTCOMES:
cardiovascular mortality | at 6 months
functional status | at 4 weeks
for the patient: NPI and ADAS-Cog | during the study
for the caregiver: ZARIT scale, questionnaire of feeling of competency, Montgomery and Asberg Depression Rating Scale (MADRS), Geriatric Depression Scale (GDS) | during the study
all cause mortality | at one year
score on a depression rating scale | at 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie Rigaud, Pr, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Assistance Publique-Hôpitaux de Paris, Paris, Île-de-France Region, France

REFERENCES:
- [Background] Wenisch E, Stoker A, Bourrellis C, Pasquet C, Gauthier E, Corcos E, Banchi MT, De Rotrou J, Rigaud AS. [A global intervention program for institutionalized demented patients]. Rev Neurol (Paris). 2005 Mar;161(3):290-8. doi: 10.1016/s0035-3787(05)85035-0. French. PMID 15800450